CLINICAL TRIAL: NCT05679895
Title: Safety and Efficacy of hCD1a-CAR T (OC-1) Therapy, in Patients With Relapsed/Refractory (R/R) T-cell Acute Lymphoblastic Leukemia/Lymphoma (T-ALL/LL
Brief Title: Safety and Efficacy of OC-1 Therapy in Patients With R/R T-ALL/LL
Acronym: CARxALL
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: OneChain Immunotherapeutics (Industry)
Collaborators: BioClever 2005 S.L. (Other); Hospital Clinic of Barcelona (Other); Hospital Sant Joan de Deu (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OC-01-21001
Record Dates: First submitted 2022-12-22; First posted 2023-01-11 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: T-cell Acute Lymphoblastic Leukemia; Lymphoblastic T-Cell Lymphoma
Keywords: CAR-T-based therapies; CD1a
MeSH Terms: conditions — Precursor T-Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental: CD1a-CAR T (Experimental): CD1a CAR T cells transduced with a lentiviral vector to express CD1a chimeric receptor domain on T cells administered with a dose-escalation approach.
  Interventions: Biological: CD1a-CAR T

INTERVENTIONS:
Biological: CD1a-CAR T — Autologous T-cells from peripheral blood, expanded and transduced with a lentivirus to express CD1a chimeric antigen receptor administered by intravenous infusion following a dose-escalation approach

SUMMARY:
First in humans, exploratory, open-label, single-arm, multicentre, non-competitive, dose escalation study to assess the safety and efficacy of CD1a-CAR T therapy in patients with relapsed/refractory (R/R) T-cell acute lymphoblastic leukemia/lymphoma (T-ALL/LL)

ELIGIBILITY:
Inclusion Criteria:

1. Children older than 2 years or adults, male and female in both groups.
2. Patients CD1a antigen blast expression ≥20% at inclusion, either immunophenotypically (flow cytometry) or histologically confirmed.
3. R/R CD1a-positive T-ALL/LL patients, including morphologic or MRD-detectable (≥1x10-4) bone marrow and/or extramedullary relapses after 2 therapy lines:

   1. Relapse after allogeneic haematopoietic stem cell transplantation (allo-HSCT)
   2. Primary refractoriness, defined as either morphologic persistence or detectable MRD (≥1x10-4) after two standard therapy lines, making the patient not candidate for allo-HSCT.
   3. Refractory first relapse.
   4. Second or further relapse.
4. Patient without reproductive capacity or else, commitment to the use of a highly effective method of contraception during the study.

Exclusion Criteria:

1. Limiting organ dysfunction, such as uncontrolled cardiac (e.g., depressed left ventricular ejection fraction (LVEF), <45%), pulmonary, liver, renal or CNS dysfunction.
2. Allo-HSCT within a timeframe <3 months, or requiring continued immunosuppressive treatment for graft versus host disease (GvHD).
3. Uncontrolled epilepsy or underlying central nervous system (CNS) severe disease.
4. Active bacterial, fungal or viral infection not controlled by adequate treatment.
5. Known HIV, active hepatitis B (HBV), or hepatitis C virus (HCV) infection.
6. Women who are pregnant (positive urine/blood pregnancy test) or lactating.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2023-01-31 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Number of adverse events grade III-IV | 1 year particularly the first 28 days after infusion
  Number of adverse events grade III-IV using common toxicity criteria (CTC)
Incidence of severe Cytokine release syndrome (CRS) and Immune effector cell-associated neurotoxicity syndrome (ICANS) | 1 year particularly the first 28 days after infusion
  Incidence of severe Cytokine release syndrome (CRS) (≥ grade III) and Immune effector cell-associated neurotoxicity syndrome (ICANS) (≥ grade II)
Non-relapse treatment-related mortality (NRM) | 1 year
  Non-relapse treatment-related mortality (NRM)
Number of adverse events of special interest (AESI) | 1 year
  Number of adverse events of special interest (AESI)
Assessment of the immunological homeostasis | 1 year
  Assessment of the immunological homeostasis, through the identification of lymphocytes subpopulations by flow cytometry at each study timepoint.
Incidence of the treatment-related dermatological events | 1 year
  Incidence of the treatment-related dermatological events
Number of patients developing dose limiting toxicity (DLT) | first 28 days after infusion
  Number of patients developing dose limiting toxicity (DLT)

SECONDARY OUTCOMES:
Remission rate | 1 year
  Percentage of patients presenting complete response (CR) or incomplete count recovery (CRi) at any point after treatment.
Response rates | 1 year
  Percentage of patients presenting CR, CRi, Complete remission duration (CRD), morphologic leukaemia-free status (MLFS), and no remission (NR).
Duration of remission | 1 year
  The duration of the remission will be assessed from the first documented date of remission status until progression (in days)
Minimal residual disease (MRD) response | 1 year
  Minimal residual disease (MRD) response by flow cytometry: blast count among patients presenting bone marrow complete response (sensitivity 10-4).
Progression-free survival (PFS) | 1 year
  time since the first OC-1 administration to the documented loss of response.
Overall survival | 1 year
  Overall survival time since first OC-1 administration to date of death.
Persistence of OC-1 | 1 year
  • Persistence of OC-1, as determined by flow cytometry and quantitative analysis by qPCR. Genomic copy number integrations of the CAR in peripheral blood (PB) T cells and percentage of CD1a CAR-expressing T cells.

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Hospital Clínic, Barcelona
  - Hospital Sant Joan de Déu, Barcelona